CLINICAL TRIAL: NCT06913400
Title: Progression of Stereopsis Recovery in Strabismic Patients: A One-Month and Three-Month Post-Surgery Evaluation
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/793
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Strabismic Amblyopia, Bilateral
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Stereopsis Recovery — This prospective longitudinal observational study aims to assess stereopsis recovery in strabismic patients at one month and three months post-corrective surgery

SUMMARY:
This prospective longitudinal observational study aims to assess stereopsis recovery in strabismic patients at one month and three months post-corrective surgery. The study will be conducted at Mayo Hospital, Lahore, and Sajjad Eye Center, Burewala, with a sample size of 34 using a purposive sampling technique. Eligible participants include patients aged ≥5 years undergoing strabismus surgery for esotropia, exotropia, or vertical deviations, with best-corrected visual acuity (BCVA) of 6/12 in both eyes. Patients with previous strabismus surgery, amblyopia, neurological conditions, or sensory strabismus will be excluded.

DETAILED DESCRIPTION:
Baseline assessments include visual acuity (Snellen Chart), ocular alignment (cover-uncover and prism cover tests), and stereopsis (Titmus Fly Test). The same tests will be repeated one month and three months post-surgery to evaluate changes. The study aims to determine whether strabismus surgery enhances binocular function and stereopsis, helping guide future treatment strategies. Data will be analyzed using paired t-tests to assess differences over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥5 years and adults) undergoing strabismus surgery for: esotropia, exotropia, vertical deviations (hypertropia or hypotropia)
* Best corrected visual acuity (BCVA) of 6/12 in both eyes
* Willingness to attend follow-up visits at 1 month and 3 months post-surgery.8

Exclusion Criteria:

* History of previous strabismus surgery
* Amblyopia
* Neurological and systemic conditions affecting vision
* Uncontrolled nystagmus and sensory strabismus
* Patients unable to complete stereopsis testing due to cognitive or physical limit

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective longitudinal observational study aims to assess stereopsis recovery in strabismic patients at one month and three months post-corrective surgery. The study will be conducted at Mayo Hospital, Lahore, and Sajjad Eye Center, Burewala, with a sample size of 34 using a purposive sampling technique. Eligible participants include patients aged ≥5 years undergoing strabismus surgery for esotropia, exotropia, or vertical deviations, with best-corrected visual acuity (BCVA) of 6/12 in both eyes.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Titmus fly test | 12 Months
  It is a contour stereo test performed at distance of 40cm. the test comprises of 3 sections:
  1. The housefly which shows large disparities and should be seen in depth by most subjects. Stereoacuity range of Random Dot Butterfly is
     * Bottom of lower wing: 1150 sec of arc
     * Tip of abdomen: 700 sec of arc
     * Top of upper wing: 2000 sec of arc
  2. There are 3 rows of animals, one animal in each row having a crossed disparity which ranges from 100, 200, 400 secs of arc.
  3. Circle patterns: this section consists of 9 patterns containing four circles. The disparities of the circles range from 800 to 40 secs of arc.

CONTACTS AND LOCATIONS:
Locations (1):
- CENUM Center Mayo Hospital Rd, Anarkali Bazaar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No